CLINICAL TRIAL: NCT00709566
Title: The Effectiveness of Exercise Therapy and Manual Therapy in Hip Osteoarthritis - A Multicentre Randomised Controlled Trial
Brief Title: EMPART - Exercise and Manual Physiotherapy Arthritis Research Trial
Acronym: EMPART
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Prof Geraldine McCarthy, Royal College of Surgeons in Ireland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RoyalCSI
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: Hip Osteoarthritis
Keywords: Hip; osteoarthritis; exercise; manual therapy
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis; Motor Activity | interventions — Exercise Therapy; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Waiting List control.
- Exercise therapy (Active Comparator)
  Interventions: Behavioral: Exercise therapy
- Combined therapy (Experimental): Combined Exercise therapy and Manual Therapy
  Interventions: Behavioral: Combined exercise and manual therapy

INTERVENTIONS:
Behavioral: Exercise therapy — Participants will attend an exercise based programme once a week for 8 weeks. This will be supplemented by a home based exercise programme.
  Arms: Exercise therapy
Behavioral: Combined exercise and manual therapy — Patients will attend physiotherapy once a week for 8 weeks, where they will receive a combination of exercise therapy and manual therapy. Exercise will be supplemented by a home based exercise programme
  Arms: Combined therapy

SUMMARY:
Hip osteoarthritis is a major cause of disability and reduced quality of life. Physiotherapy, which encompasses a range of interventions such as exercise therapy, manual therapy, education and electrophysical agents, is a core component of management. To date, exercise therapy to date has the greatest evidence of effect . However, this evidence is limited as only a short-term benefit has been identified and improvements in pain and function decline over time. There is some limited evidence for a beneficial effect of manual therapy over exercise. However, clinically these interventions are used in combination, not in isolation. To date, no research has investigated the combined effect of exercise and manual therapy in hip OA.

A multi-centre randomised controlled trial that compares the clinical effectiveness of a combination of manual therapy and exercise to exercise therapy only will be conducted.

DETAILED DESCRIPTION:
A multi-centre RCT that evaluates the clinical effectiveness of two physiotherapy interventions for patients with osteoarthritis of the hip will be conducted The methodology will follow CONSORT (Consolidation of Standards of Reporting Trials) guidelines. Ethical approval for the study has been obtained from the Research Ethics Committees of the participating hospitals (Beaumont, St Vincent's University, Mater Misercordiae University Hospitals, Adelaide Meath Hospital Dublin, incorporating National Children's Hospital). Patients will be assessed at baseline, 9 weeks, (end of treatment) and 18 weeks. The treating therapists will be blinded to outcome assessments. Subjects cannot be blinded due to the nature of the interventions.

All patients with a diagnosis of Hip OA referred for physiotherapy from rheumatologists, GPs and orthopaedic consultants will be considered for inclusion into the RCT. Four similarly matched physiotherapy departments will be used: Beaumont Hospital (BH), St Vincent's University Hospital (SVUH) Adelaide Meath Hospital Dublin, incorporating National Children's Hospital) and Mater Misericordiae University Hospital (MMH).

Consenting subjects will be randomly allocated to one of 3 groups

1. Exercise therapy (comprising strengthening, range of motion and aerobic exercise)
2. Combined Exercise therapy and Manual Therapy
3. Control group (Waiting List). These patients will remain on the waiting list for a 9 week period and will then be randomized to one of the two intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Clinical criteria for the diagnosis of hip osteoarthritis (American College Rheumatology) (Altman et al, 1991):

  * Subjective complaint of hip pain with either hip internal rotation < 15 degrees and hip flexion <115 degrees or >15 degrees hip internal rotation and pain on hip internal rotation
  * morning stiffness less than or equal to 60 minutes, age > 50 years.
* Age 40-80 years except in 2 above (age >50 years).
* Radiological evidence of osteoarthritis (2 of the following 3 criteria):

  * osteophytes
  * joint space narrowing
  * ESR<20mm/hr (American College of Rheumatology Criteria for the Classification and Reporting of Osteoarthritis of the Hip)
* Referred for physiotherapy

Exclusion Criteria:

* Previous hip arthroplasty, history of congenital/adolescent hip disease
* Clinical signs of lumbar spine disease
* Physiotherapy in previous 6 months
* Pregnancy
* Hip fracture
* Contraindications to exercise therapy
* Contraindications to manual therapy
* On waiting list for joint replacement within the next 18 weeks
* Rheumatic diseases e.g. Rheumatoid Arthritis, Ankylosing Spondylitis, etc
* Hip cortisone injection in previous 30 days

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
WOMAC (Western Ontario and McMaster Universities) Osteoarthritis Index Physical Function Subscale | 0, 9, 18 weeks

SECONDARY OUTCOMES:
Numerical Rating Scale for Pain | 0,9,18 weeks
WOMAC total score, pain and stiffness subscales | 0,9,18 weeks
Global Assessment of Change- 7 Point Likert Scale | 9,18 weeks
Hip Range of motion using goniometry | 0,9,18 weeks
Short Form-36v2 (Quality of Life) | 0,9,18 weeks
Hospital Anxiety and Depression Scale (HADS) | 0,9,18 weeks
Physiotherapy Out-Patient Survey for Patient Satisfaction | 18 weeks
Medication Usage (pain diary and Medication Quantification Scale) | 0,9,18 weeks
International Physical Activity Questionnaire (Short version) | 0,9,18 weeks
Repeated sit to stand test | 0,9,18 weeks
50 foot walk test | 0,9,18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine McCarthy, MD, FRCPI, Principal Investigator — Royal College of Surgeons in Ireland; Tara Cusack, PhD, Principal Investigator — University College Dublin, Ireland; Helen French, MSc, Principal Investigator — Royal College of Surgeons in Ireland
Locations (4):
- Ireland (4):
  - Adelaide Meath Hospital Dublin incorporating the National Childrens Hospital, Dublin, Dublin
  - St Vincent's University Hospital, Dublin, Dublin
  - Mater Misericordiae University Hospital, Dublin, Dublin
  - Beaumont Hospital, Dublin, Dublin

REFERENCES:
- [Background] French HP (2007). Physiotherapy management of osteoarthritis of the hip: a survey of current practice in acute hospitals and private practice in the Republic of Ireland, Physiotherapy, 93 (4), 253-260.
- [Background] French HP, Cusack T, Brennan A, White B, Gilsenan C, Fitzpatrick M, O'Connell P, Kane D, Fitzgerald O, McCarthy GM. Exercise and manual physiotherapy arthritis research trial (EMPART): a multicentre randomised controlled trial. BMC Musculoskelet Disord. 2009 Jan 19;10:9. doi: 10.1186/1471-2474-10-9. PMID 19152689